CLINICAL TRIAL: NCT05065008
Title: Investigate the Roles of Gut Microbiome in the Differential Responses of UTI Susceptible Women to Cranberry Juice Intake
Brief Title: The Roles of Gut Microbiome in UTI Susceptible Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09003; IRB202102165 (Other: UF IRB-01); PRO00039868 (Other: UF UFIRST)
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Cranberry; UTI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranberry juice consumption (Experimental): Participants deemed as responders and non-responders will be given 20-30 oz (590-885 mL) of cranberry juice daily for 3 weeks.
  Interventions: Other: Cranberry juice
- Apple juice consumption (Experimental): Participants deemed as responders and non-responders will be given 20-30 oz (590-885 mL) apple juice with matching sugar and calories daily for 3 weeks.
  Interventions: Other: Apple juice

INTERVENTIONS:
Other: Cranberry juice — The responders and non-responders will drink 20-30 oz of (590-885 mL) 27% cranberry juice daily for 3 weeks.
  Arms: Cranberry juice consumption
Other: Apple juice — The participants will drink apple juice with matching sugar content and calories for 3 weeks
  Arms: Apple juice consumption

SUMMARY:
Clinical trials on cranberry juice and UTI prevention yielded both positive and negative results for unknown reason. Gut microbiome in women affect the absorption and metabolism of cranberry bioactives. The variation of gut microbiome is a probable mechanism for metabolic polymorphisms and disparity in UTI prevention in women.

DETAILED DESCRIPTION:
The American cranberries, especially cranberry juice, have used for centuries as a folk medicine to prevent urinary tract infections (UTI), which affect 50% of women in their lifetime. Over 40 clinical trials have been conducted in the last 20 years to verify the UTI preventatively activity of cranberry juices, but the results were contradictory. About 90% of UTI are initiated by the adhesion of uropathogenic E. coli (UPEC) on urinary tract epithelia. It was reported that human urine after consumption of cranberry juice inhibited the adhesion of UPEC. The A-type proanthocyanidins and xyloglucans are the presumed bioactives in cranberries, however, this is unlikely because these two classes of compounds have extremely low bioavailability in human body. Preliminary research suggested that women can be either "resistant" or "susceptible" to UTI depending on the inherent anti-adhesion activity in their urine against UPEC before consuming cranberry juice. Not all but a fraction of "UTI susceptible" women had increased urinary anti-adhesion activity after consuming cranberry juices. These women are classified as "responders" and others are "non-responders". The variation of gut microbiome is a probable mechanism for metabolic polymorphisms and disparity in UTI prevention. The objective of this trials is to identify gut microbes and anti-adhesive urinary biomarkers which significantly contribute to the anti-adhesion of UPEC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women participants;
* BMI 18.5-29.9 kg/m2;
* At least 110 pounds in weight

Exclusion Criteria:

* BMI≥ 30 kg/m2;
* Pregnancy and breast-feeding;
* Smoking, frequent alcohol use;
* History of any clinically important disorder that may interfere with interpretation of the results;
* Intake of medication that might influence the outcome of the study

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women is a group which is susceptible to urinary tract infections (UTIs) based on previous papers. This study will determine American cranberries to prevent UTIs in susceptible women.
Enrollment: 160 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in the unrinary anti-adhesion activity of UTI susceptible women | Baseline up to 21 days of each intervention
  Compare the statistical differences between the changes from baseline in the an-adhesion activity against uropathogenic E. coli in UTI-susceptible women after consuming the cranberry juice for 3 weeks versus after consuming the placebo juice for 3 weeks. Anti-adhesion activity in urine will be measured using a fluorescence-based microplate method. The anti-adhesion activities of urines will be expressed by its equivalence to myricetin level. The unit for urine anti-adhesion activities is µg myricetin/mg creatinine.

SECONDARY OUTCOMES:
Determine the compositional differences of gut microbiome in responders and non-responders after the cranberry juice intake | Baseline up to 21 days of each intervention
  Compare the differences in the gut microbiomes between responders and non-responders after consuming the cranberry juice for 3 weeks versus after consuming the placebo juice for 3 weeks. Human feces collected from responders and non-responders will be analyzed for microbiota composition. Relative abundance of gut microbiome at phylum level, family level, genus level, and Firmicutes over Bacteroidetes ratio will be evaluated. Genomic microbial DNA will be extracted from fecal samples using DNA isolation kits. The 16S ribosomal RNA gene (V1-3 region) of each sample will be amplified and sequenced using a barcoding system on a MiSeq sequencer. Sequence data will be analyzed using the latest version of QIIME.
Identify anti-adhesion urinary biomarkers in responders versus non-responders after the cranberry juice intake | Baseline upt to 21 days of each intervention
  Determine the impacts of cranberry juice intake on the urinary metabolome and identify anti-adhesion urinary biomarkers in responders and non-responders after consuming the cranberry juice for 3 weeks versus after consuming the placebo juice for 3 weeks. Metabolites in urine will be detected using UHPLC-HRMS and annotated using combination of m/z and retention time. Metabolites that significantly contribute to the anti-adhesion activity of urine revealed by PLS regression analysis are the potential anti-adhesion biomarkers. A list of potential biomarkers will be generated. Structures of these biomarkers will be tentatively determined through spectral analysis and database searching. Structure of tentatively identified biomarkers will be confirmed by comparing with authentic standards.

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Gu, PhD, Principal Investigator — University of Florida; Gary P Wang, PhD, Study Director — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States